CLINICAL TRIAL: NCT04494464
Title: Awareness, Treatment Rates and Compliance to Treatment in Patients With Serum LDL Cholesterol Higher Than 250 mg/dL, and Possible, Probable or Definite Familial Hypercholesterolemia
Brief Title: Treatment Rates and Compliance to Treatment in Patients With Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Didem Ozdemir, Clinical Professor, Ankara Yildirim Beyazıt University
Other Study IDs: Hypercholesterolemia
Record Dates: First submitted 2020-07-24; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with LDL cholesterol ≥250 mg/dL: Patients older than 18 years old and have a serum LDL-C≥250 mg/dL between January 2010 and December 2016. Patients with a serum TSH≥10 mIU/mL, patients with glomerulonephritis or nephrotic syndrome, patients with ALT or AST higher than 3 times of normal limits and patients with serum triglyceride >400 mg/dL were excluded.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Familial hypercholesterolemia is a genetic disease characterized by increased levels of low density lipoprotein cholesterol (LDL-C). It is underdiagnosed and undertreated despite relatively high prevalence and significant association with increased mortality.

DETAILED DESCRIPTION:
Patients older than 18 years old and have a serum low density LDL-C≥250 mg/dL were identified from the hospital database. A questionnaire was completed via phone. Patients were classified as definite, probable and possible familial hypercholesterolemia according to Dutch Lipid Clinical Network Criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old and have a serum LDL-C≥250 mg/dL

Exclusion Criteria:

* Patients who refuse dto interview
* Serum TSH≥10 mIU/mL
* Glomerulonephritis or nephrotic syndrome
* ALT or AST higher than 3 times of normal limits
* Serum triglyceride >400 mg/dL

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old and have a serum LDL-C≥250 mg/dL
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Treatment rates | January 2010 and December 2016
  Patients with a serum LDL-C≥250 mg/dL were identified from the database of our hospital. Dutch Lipid Clinical Network Criteria was used to classify patients as definite, probable and possible FH. Patients were reached by phone and a questionnaire was applied. The questionnaire consisted of questions related with clinical and physical examination findings defined in theDutch Lipid Clinical Network Criteria. Total cholesterol, LDL-C, HDL-C, triglyceride levels were obtained from the medical records. Patients were asked whether they were using lipid lowering drugs. If they were not using, the cause of this was asked. By this way, we determined the rate of use of lipid lowering drugs in patients with LDL-C≥250 mg/dL and have definite, probable or possible familial hypercholesterolemia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaman S, Ozdemir D, Akman BT, Cakir B, Ersoy O. Awareness, treatment rates, and compliance to treatment in patients with serum LDL cholesterol higher than 250 mg/dL, and possible, probable, or definite familial hypercholesterolemia. Postgrad Med. 2021 Mar;133(2):146-153. doi: 10.1080/00325481.2020.1805212. Epub 2020 Sep 23. PMID 32744105